CLINICAL TRIAL: NCT02578004
Title: Case Control Study of the Risk Factors for Pressure Ulcers in Tunisian Patients
Brief Title: Risk Factors for Pressure Ulcers
Status: Completed | Type: Observational
Sponsor: Centre Hôpital Universitaire Farhat Hached (Other)
Responsible Party: Principal Investigator, latifa, PhD, Centre Hôpital Universitaire Farhat Hached
Other Study IDs: CHU Farhat Hached
Record Dates: First submitted 2015-10-09; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Pressure Ulcers
Keywords: Difficult; environmental, microbial, immunological and genetic factors; significantly different
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 100 patients suffering from pressure ulcer: 100 subjects were having at least one wound of pressure ulcer (74 men and 26 women) middle-aged (55.5±20 years) and were recruited from many services of three University Regional hospitals of Tunisia.
  Interventions: Other: biochemical and molecular analysis
- 213 healthy subjects: 213 healthy subjects (125 men and 88 women) middle-aged (51.5±17 years). Although, healthy individuals, were included as controls, followed in the outpatient services of the University Hospital Farhat Hached and they considered clinically free of pressure ulcer and tissue necrosis.
  Interventions: Other: biochemical and molecular analysis

INTERVENTIONS:
Other: biochemical and molecular analysis

SUMMARY:
Development of pressure ulcer (PU) is complex and multifactorial. The association of a constituted PU and of clinical / biological major elements is demonstrated and justifies. Prevention of PU is an important health priority, one that requires clear identification of risk factors.

ELIGIBILITY:
Inclusion Criteria:

* presenting with at least of a wound and confirmed diagnosis of PU, age≥18 years old, bedridden, not feeds only and without trophic and mental disorders.

Exclusion Criteria:

* paediatric study populations, age > 90 years old, allergy to wound products, malignant origin

Ages: 19 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective study consisted of 100 patients were having at least one wound of pressure ulcer that met the following inclusion criteria. Who followed in many departments (emergency, orthopedic, physical medicine) of three University Regional hospitals of Tunisia (Farhat Hached and Sahloul Sousse, Fattouma Bourguiba Monastir) were evaluated prospectively.
Sampling Method: Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2013-01; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Anthropometric characteristics | one hour
  Body Mass Index (BMI) is a simple index of weight-for-height. It is defined as the weight in kilograms divided by the square of the height in metres (kg/m2).
Diabetes mellitus | one hour
  - Plasma levels glucose in mmol/l was measured by standard enzymatic methods using reagents in a fully automated analyzer Cx5 Pro-Bechman Coulter-Fuller-Ton
Dyslipidemia | one hour
  * Lipid markers: total serum cholesterol (CH), serum triglyceride, serum HDL- CH, in mmol/l, levels were measured by standard enzymatic methods using reagents in a fully automated analyzer (Randox Antrim, UK; CX9-BECKMANN).
  * Low density lipoprotein cholesterol (LDL-C) in mmol / l was determined by Friedewald formula.
  * non esterified fatty acids in serum was determined by colorimetric method at 550 nm (mmol/l)
Renal failure | one hour
  - renal profile: urea (mmol/l), creatinine and uric acid (μmol/l) levels were measured by standard enzymatic methods using reagents in a fully automated analyzer ( Cx9 Pro-Bechman Coulter-Fuller-Ton).
Inflammatory parameter | one hour
  - C-reactive protein (CRP), in mg/l, was measured using immunoturbidimetric methods (COBAS INTEGRA 400 Roche).
Endogenous inflammatory marker | one hour
  - α1-acid glycoprotein, in g/l, measured using the dry chemistry method (BN prospec, siemens)
Markers of nutritional status | one hour
  * albumin (chronic marker) and prealbumin (early marker) were measured, in g/l, using the dry chemistry method (BN prospec, siemens).
  * Protide in g/l was measured by standard enzymatic methods using reagents in a fully automated analyzer (CX9-BECKMANN).
Marker of lipid peroxidation | one day
  * Serum total homocysteine concentrations in μmol/l were measured by using an AxSYM (ABBOTT) homocysteine assay.
  * thiobarbituric acid reactive substances (TBARS) in serum was determined by the fluorimetric method of Yagi in μmol/l.
Antioxidant parameters | one day
  - Serum catalase activity in KU/l was determined according to the spectrophotometric method of Goth .
Total antioxidant status | one hour
  Serum total antioxidant status in mmol/l was measured with RANDOX kit (Cat. No. NZ 2332; Randox Labs Ltd., Crumlin, UK) by colorimetric method at 600 nm .
Determination of trace elements | one hour
  Serum copper in μmol/l was indicated spectrophotometrically with RANDOX kit (Cat. No. CU 2340; Randox Labs Ltd., Crumlin, UK) at 580 nm according.
  Serum zinc was measured in μmol/l with RANDOX kit (Cat. No. ZN 2341; Randox Labs Ltd, Crumlin, UK) at 560 nm.
Nutritional status | 3 hours
  - Nutritional Risk Index (NRI) was originally derived from the serum albumin concentration and the ratio of present to usual weight [NRI = (1.489 x albumin, g/L) + (41.7 x present weight/ideal body weight)] and categorized as follows: severe risk (NRI < 83.5), moderate risk (83.5 < NRI < 97.5) and no risk (NRI > 97.5).
Nutritional risk | 3 hours
  - Prognostic Inflammatory and Nutritional Index (PINI) is a simple clinical [PINI = AAG x CRP / albumine x prealbumin] and classificated as follows: normal (1<PINI score <10), mild malnutrition (11<PINI score<20), severe malnutrition (21<PINI score<30) and risk for death when PINI score >30.
  These scores gained in popularity as it uses an objective rather than subjective measurements to determine nutritional risk in hospitalized patient populations.
A microbiological diagnosis | 3 days
  The bacterial colonization of a wound is a recognized detrimental factor in the multifactorial process of wound healing.
  wound per patient suffering from pressure ulcer was cultured by swab to determine the bacterial species of the infection and helps guide antibiotic therapy.
  The representative sample is collected before topical or systemic antibiotics are initiated and pain assessment should be conducted prior to wound procedures such as dressing changes and debridement. Bacterial swabs provide information on the predominant flora.
Proteomics | 2 days
  - Serum gelatinase activities of MMP-9 by zymography (%)
DNA extraction | 2 days
  Genomic DNA was extracted from whole blood using the salting out method for the part of molecular biology.
Genotype for the MMP9-1562 C/T polymorphism | 1 days
  * Genetic polymorphism in the MMP9 coding region 1562C>T was screened following the polymerase chain reaction and restriction fragment length polymorphism (RFLP-PCR).
  * The frequency distributions of different MMP9-1562 C/T genotypes and allele were investigated.
  * The relationship between the polymorphism of the MMP-9 gene and the severity of PU was analyzed.
Genotyping of TNF- α G238A | 1 days
  * TNF-α G238A promoter polymorphism were determined by the RFLP-PCR method.
  * The genotypic and allelic frequencies of -238G/A were calculated
  * This study investigated the association between TNF-α-238G>A and Pressure ulcer in Tunisian population.
Genotyping of TNF- α G308A | 1 days
  * The genotypic analysis of the TNF-α G308A polymorphism was performed using Allele-specific PCR (AS-PCR) amplification.
  * In this study, we have analyzed the TNF-α gene promoter -308G/A polymorphism in Tunisian patients with PU to evaluate the contribution of this SNP in genetic susceptibility to PU.

CONTACTS AND LOCATIONS:
Locations (1):
- Latifa KHLIFI, Sousse, Tunisia